CLINICAL TRIAL: NCT03304418
Title: A Phase 2 Study of Radium-223 and Radiotherapy in Hormone-Naïve Men With Oligometastatic Prostate Cancer to Bone
Brief Title: Radium-223 and Radiotherapy in Hormone-Naïve Men With Oligometastatic Prostate Cancer to Bone
Acronym: RROPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI102312
Record Dates: First submitted 2017-09-27; First posted 2017-10-09 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer Metastatic to Bone
MeSH Terms: interventions — radium Ra 223 dichloride; Radiation

STUDY DESIGN:
Intervention Model Description: This is a phase IIa, open label, single arm, prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radium Ra 223 dichloride and radiation, all patients (Experimental)
  Interventions: Drug: Radium Ra 223 Dichloride; Radiation: Radiation

INTERVENTIONS:
Drug: Radium Ra 223 Dichloride — Radium Ra 223 dichloride will be delivered intravenously at 55 kBq/kg (1.49 mCi)/kg (+/- 10% total dose) for a total of six cycles. 1 cycle= 28 days. The first cycle will commence at study enrollment, then cycles 2-6 will commence after the completion of radiotherapies at 4 week intervals
  Other Names: Xofigo
Radiation: Radiation — All external beam radiations oligometastatic sites will commence after cycle 1 of Radium-223 but prior to cycle 2 of Radium-223. All subjects will receive Stereotactic body or hypofractionated radiation to sites of bone disease seen on imaging studies. Patients will have the primary tumor sites and 5 or fewer sites of bone-only metastasis treated with external beam radiation.
  Any of the following regimens are considered ablative, acceptable and are biologically equivalent to 60Gy EQD2:
  * Single fraction: 16 Gy total at 16 Gy per fraction (SBRT)
  * Three fractions: 24 Gy total at 8 Gy per fraction (SBRT)
  * Five fractions: 30 Gy total at 6Gy per fraction (SBRT).When using five fractions, can reduce to 25 Gy total at 5 Gy per fraction (SBRT) or to a minimum of 20 Gy total at 4 Gy per fraction (SBRT), per treating investigator.
  * Six fractions: 32.4 Gy total at 5.4Gy per fraction (Hypofractionated)

SUMMARY:
This is a phase IIa, open label, single arm, and prospective study of hormone therapy-naïve men with oligometastatic prostate cancer to the bone. The study will test if treating the primary tumor sites and 5 or fewer sites of bone-only metastasis with external beam radiation with concomitant systemic Radium-223 will reduce the utilization of androgen deprivation therapy, improve QOL and improve OS over a the comparator cohort of SWOG intermittent ADT historic cohort.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic or symptomatic hormone naïve men with testosterone levels ≥100 ng/dL with previously treated localized prostate cancer who now have rising PSA's and five or fewer bone metastases.
* Subjects who have been previously treated with definitive and/or adjuvant/salvage radiotherapy to the primary site and/or regional lymph nodes with concurrent ADT are allowed if the last hormone therapy delivered > 6 months prior. Subjects who have had more than 30 days and fewer than 45 days of bicalutamide monotherapy for any reason within the 6 months prior to enrollment are eligible for the study, providing they have been off of the drug for at least 30 days prior to enrollment. Subjects who have had fewer than 30 days of bicalutamide are eligible for the study, as long as they discontinue the drug at least 5 days prior to the first study treatment.
* Histologic confirmation of Prostate Adenocarcinoma diagnosis.
* Age ≥ 18 years.
* Life expectancy of at least 2 years.
* Acceptable hematology and serum biochemistry screening values:

  * White Blood Cell Count (WBC) ≥ 3,000/mm3
  * Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
  * Platelet (PLT) count ≥ 100,000/mm3
  * Hemoglobin (HGB) ≥ 10 g/dl
  * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Creatinine ≤ 1.5 x ULN
  * Albumin > 2.5 mg/dL
* Willing and able to comply with the protocol, including follow-up visits and examinations.
* Karnofsky Performance Score >60 or ECOG equivalent.
* Radiographic confirmation of oligometastatic diagnosis via Bone Scan validated by either CT scan or MRI or PET/CT with Fluciclovine within the past 90 days.
* Subjects who have not had surgical removal of their prostate and have a partner of child bearing potential must agree to use condoms beginning at the signing of the ICF until at least 6 months after the last dose of study drug. Because of the potential side effect on spermatogenesis associated with radiation, female partners of childbearing potential must agree to use a highly effective contraceptive method during and for 6 months after completing treatment
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Men with known brain or visceral metastases (except regional lymph nodes as defined by section 5.2.5) defined by CT or MRI Imaging of the abdomen or pelvis.
* Men who have had LHRH agonist or antagonist hormone therapy in the prior six months.
* Men with >5 bony metastases.
* Men with baseline serum Testosterone <100 ng/dL.
* Men with new or progressing lymphadenopathy clearly consistent with prostate metastasis on imaging or proven by pathologic biopsy at any time three months or later following their initial definitive therapy.
* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 3 years. All patients with in situ carcinoma are eligible for this study (for example, carcinoma in situ of the oral cavity is eligible) except patients with carcinoma of the bladder (including in situ bladder cancer or superficial bladder cancer).
* Use of finasteride within 30 days prior to therapy PSA should not be obtained prior to 30 days after stopping finasteride.
* Use of dutasteride within 90 days prior to therapy. PSA should not be obtained prior to 90 days after stopping dutasteride.
* Previous or concurrent cytotoxic chemotherapy for prostate cancer.
* Received systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or Radium Ra 223 dichloride) for the treatment of bony metastases.
* Men who will receive radical prostatectomy to the primary site.
* Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Spinal Cord compression will be defined as 360 degree circumferential obliteration of T2 cerebrospinal fluid signal around the spinal cord. Treatment should be completed for spinal cord compression.
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol. (Patients on Coumadin or other blood thinning agents are eligible for this study.)
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
* Cardiac failure New York Heart Association (NYHA) III or IV Crohn's disease or ulcerative colitis.
* Bone marrow dysplasia.
* Fecal incontinence.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Radium Ra 223 Dichloride and Radiation, All Patients: Radium Ra 223 Dichloride: Radium Ra 223 dichloride will be delivered intravenously at 55 kBq/kg (1.49 mCi)/kg (+/- 10% total dose) for a total of six cycles. 1 cycle= 28 days. The first cycle will commence at study enrollment, then cycles 2-6 will commence after the completion of radiotherapies at 4 week intervals
  Radiation: All external beam radiations oligometastatic sites will commence after cycle 1 of Radium-223 but prior to cycle 2 of Radium-223. All subjects will receive Stereotactic body or hypofractionated radiation to sites of bone disease seen on imaging studies. Patients will have the primary tumor sites and 5 or fewer sites of bone-only metastasis treated with external beam radiation.
  Any of the following regimens are considered ablative, acceptable and are biologically equivalent to 60Gy EQD2:
  * Single fraction: 16 Gy total at 16 Gy per fraction (SBRT)
  * Three fractions: 24 Gy total at 8 Gy per fraction (SBRT)
  * Five fractions: 30 Gy total at 6Gy per fraction (SBRT).When using five fractions, can reduce to 25 Gy total at 5 Gy per fraction (SBRT) or to a minimum of 20 Gy total at 4 Gy per fraction (SBRT), per treating investigator.
  * Six fractions: 32.4 Gy total at 5.4Gy per fraction (Hypofractionated)
Period: Overall Study
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Requiring Androgen Deprivation Therapy (ADT) Use at 15 Months
Description: To determine if 20% of ADT naïve men treated with concurrent EBRT and Radium-223 will not require ADT for progression by 15 months.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Number analyzed (Participants) | 20
Participants | 10

2. Secondary Outcome: Median Time From Start of Study Therapy to Start of ADT
Description: Determine the hormone-therapy free survival time for men treated with concurrent EBRT and Radium-223 and determine if it is a 30% risk reduction over the SWOG intermittent ADT historic cohort
Time Frame: 2 years
Population: 8 of 20 total patients did not begin ADT while on study, so 12 of 20 patients were evaluated for this measure
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Number analyzed (Participants) | 12
Days | 260 (200.2)

3. Secondary Outcome: Mean Expanded Prostate Inventory Composite (EPIC) Scores at End of Treatment
Description: To evaluate health related quality of life (QOL) as scored by the 50 item Expanded Prostate Inventory Composite (EPIC) EPIC urinary, bowel, sexual and hormonal domains.
  EPIC assesses the disease-specific aspects of prostate cancer and its therapies and comprises four summary domains (Urinary, Bowel, Sexual and Hormonal). Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health-related quality of life.
Time Frame: 6 months
Population: Of the 20 total participants, 10 completed the EPIC questionnaire at the End of Treatment timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Number analyzed (Participants) | 10
score on a scale
  Urinary Summary Score | 74.1 (17.8)
  Bowel Summary Score | 89.1 (10.9)
  Sexual Summary Score | 12.4 (9.8)
  Hormonal Summary Score | 81.9 (17.5)

4. Secondary Outcome: Mean PROMIS-29 Scores at End of Treatment
Description: To evaluate health related quality of life (QOL). The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) will be used to assess general function and well-being.
  The raw score for each PROMIS instrument is converted to a T-score on a scale of 0-100. For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10. A higher PROMIS T score represents more of the concept being measured. For negatively worded concepts like Anxiety, a T score of 60 is one SD worse than average. By comparison, an Anxiety T score of 40 is one SD better than average. However, for positively worded concepts like Physical Function Mobility, a T score of 60 is one SD better than average while a T score of 40 is one SD worse than average.
Time Frame: 6 months
Population: Of the 20 total participants, 10 completed the EPIC questionnaire at the End of Treatment timepoint
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Number analyzed (Participants) | 10
T-scores
  Pain Interference | 53.5 (9.3)
  Depression/Sadness | 44.7 (6.1)
  Physical Function | 46.9 (11.2)
  Fatigue | 47 (10.1)
  Anxiety/Fear | 45.2 (6.6)
  Sleep Disturbance | 49.1 (7.7)
  Satisfaction with Social Roles and Activities | 49.8 (7.7)

5. Secondary Outcome: Evaluate Time to First Skeletal Related Event (SRE)
Description: Documentation of complications associated with bone metastases and may include (but not limited to) fractures, spinal cord compression, bone pain, and hypercalcemia.
Time Frame: 2 years
Population: Of 20 evaluable participants, two experienced a skeletal related event.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Number analyzed (Participants) | 2
Days | 554.5 (154.9)

6. Secondary Outcome: Evaluate the PSA Doubling Time
Description: This outcome measure will report the mean time elapsed from baseline PSA to PSA to double in value. Participants were followed for 24 months from the initiation of study treatment. PSA doubling time was censored at 24 months.
Time Frame: 2 years, assessed at every visit in that time period
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Number analyzed (Participants) | 20
months | 19.32 (8.26)

7. Secondary Outcome: Evaluate Overall Surival
Description: This outcome measure will report the overall survival at 2 years. Patients were followed for survival for two years after study enrollment. Patients who refused follow-up were censored at their off-study date.
Time Frame: 2 years after study enrollment
Measure: Mean (Standard Deviation); unit: month
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
Number analyzed (Participants) | 20
month | 22.98 (4.55)

ADVERSE EVENTS:
Time Frame: The collection of all adverse events will begin after the first dose of study treatment and end 30 days after the last dose of study treatment. The collection of treatment-related adverse events will continue until the last study visit (or until new cancer treatment is initiated, if sooner).
Arm/Group | Radium Ra 223 Dichloride and Radiation, All Patients
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium Ra 223 Dichloride and Radiation, All Patients (N=20)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium Ra 223 Dichloride and Radiation, All Patients (N=20)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 14 (16)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03304418/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03304418/ICF_004.pdf